CLINICAL TRIAL: NCT06173479
Title: Effect of a Health Belief Model-Based Educational Intervention (HeBSaPU) on Safe Pesticide Use Practices and Biomarkers in Greenhouse Agriculture Workers in Antalya, Turkey
Brief Title: Health Belief Model-Based Educational Intervention on Safe Pesticide Use and Biomarkers in Agricultural Workers
Acronym: HeBSaPU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dilek AYAZ (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Dilek AYAZ, M.Sc., Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RCT829741
Record Dates: First submitted 2023-12-05; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Exposure Occupational; Safety Issues; Health Behavior; Nurse's Role
Keywords: greenhouse agricultural workers; pesticide exposure; health belief model; educational interventions
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: randomized controlled, single-blind experimental design with a pretest-posttest control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HeBSaPU (Experimental): HeBSaPU is an acronym for educational interventions for safe pesticide use based on the health belief model. The HeBSaPU arm will get interventions for 12 weeks. HeBSaPU include educational posters, free personal protective equipment (PPE) incentives, reminder short messages, and demonstration components about correct PPE usage.
  Interventions: Behavioral: HeBSaPU
- Control (Active Comparator): The control arm will not take any interventions.
  Interventions: Behavioral: HeBSaPU

INTERVENTIONS:
Behavioral: HeBSaPU — HeBSaPU training content explains the definition of pesticides, their way of entry into the body, and their health effects. Personal protective equipment, personal hygiene behaviors, and safe behaviors regarding the correct and safe use of pesticides were mentioned.

SUMMARY:
Brief Summary:

Purpose: This clinical trial aims to investigate the effect of educational interventions (HeBSaPU) based on the Health Belief Model on safe pesticide use and biomarkers among greenhouse agricultural workers. The main questions it aims to answer are;

1. Compared to the control group, HeBSaPU affects safe pesticide use practices in greenhouse agricultural workers.
2. Compared to the control group, HeBSaPU affects safe pesticide use health beliefs in greenhouse agricultural workers.
3. Compared to the control group, HeBSaPU affects pesticide exposure determined by urine samples in greenhouse agricultural workers.

Participants took educational interventions based on Health Belief Model (HBM) sub-dimensions; including educational posters, free personal protective equipment (PPE) incentives, short reminder messages, and demonstration components about correct PPE usage.

DETAILED DESCRIPTION:
The study aims to determine the effect of Health Belief Model (HBM) based educational interventions on safe pesticide use practices and biomarkers in greenhouse agricultural workers in Antalya, Turkey.

This research is a single-blind (participants), superiority randomized controlled trial design with a parallel group. The population of the research will be the greenhouse agricultural workers in the Sarıcasu Village of Antalya Province. In determining the research sample, the "effect of educational interventions on the change in protection behavior" was taken as Hegges g=0.89, and the sample number was calculated as 56 individuals with a 5% type 1 error margin. Considering that there would be losses during the research, it was planned to take 15-20% more of the sample (n=66).

On the map obtained from the Geographical Information Systems of Sarıcasu village, the greenhouses were randomized as experimental and control groups with the help of Randomizer.org.

Safe Pesticide Use Practices questionnaire, and Safe Pesticide Use Behaviors Health Belief Model Scale will be used to collect data. The variation of individuals' pesticide exposures will be determined by residue determination in urine samples.

Pre-testing of the study, taking the first urine samples, and starting the educational interventions will take place in the second week of November. At the end of twelve weeks, it is anticipated that the data collection process will be terminated with the collection of the last tests and the second urine samples in the last week of January.

At the end of the research, it is expected that the safe pesticide use behaviors of HBM-based education initiatives will change positively, and the diacyl phosphate metabolite concentrations in the urine will decrease with the effect of this change.

ELIGIBILITY:
Participant inclusion criteria

* Age: 18-65 years, inclusive
* Being a greenhouse agricultural worker
* Being a permanent employee in pesticide-related jobs in selected greenhouses,
* No communication-related barriers (language, speaking, understanding, etc.)
* Volunteering to participate in research

Participant exclusion criteria

* Being a seasonal agricultural worker
* Being a daily wage worker,
* Not dealing with pesticide-related works

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-01-28 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Dialkylphosphates metabolites in urine samples | For 12-weeks
  The concentration of four metabolites (Dimethyl phosphate, Diethyl phosphate, O,O-Dimethyl Dithiophosphate, O,O-Diethyl Dithiophosphate) is expected to change in urine samples.
Safe Pesticide Use Practice Level | For 12-weeks
  Safe Pesticide Use Practice Questionare: A minimum of 20 and a maximum of 100 points are obtained from the questionnaire. A higher total score means a higher pesticide safety level.
Health Beliefs for Safe Pesticide Use Practices | For 12-weeks
  Health Belief Model Scale for Safe Pesticide Use Practices: A minimum of 39 and a maximum of 195 points are obtained from the scale. An increase obtained from the scale is interpreted as a positive health belief level.

CONTACTS AND LOCATIONS:
Overall Officials: Dilan Akın, Study Chair — The Scientific and Technological Research Council of Turkey
Locations (1):
- Akdeniz University, Antalya, Konyaaltı, Turkey (Türkiye)